# Statistical Analysis Plan

| TRIAL FULL TITLE | Doravirine concentrations and antiviral activity in genital fluids in HIV-1 infected individuals ("DORAGEN Study") |
|---|---|
| SAP VERSION | 1.0 |
| SAP VERSION DATE | 06/05/2019 |
| Protocol Version (SAP associated with) | 1.2 |

## **Principal Investigator**

Daniel Podzamczer, M.D, PhD.

HIV and STD Unit -Infectious Diseases Department

Hospital Universitari de Bellvitge

### **Author**

Antonio Navarro, MSc

HIV and STD Unit -Infectious Diseases Department

Hospital Universitari de Bellvitge

**Protocol identification number: DORAGEN** 

ClinicalTrials.gov Identificator: NCT04097925

Signature page

Principal investigator:

Daniel Podzamczer (06/05/2019)

**Author:** 

Antonio Navarro (06/05/2019)

## **Abbreviations**

HIV Human Immunodeficiency Virus

TAF Tenofovir Alafenamide Fumarate

FTC Emtricitabine

ART Antirretroviral Treatment

PK Pharmacokinetics

PD Pharmacodynamics

# Table of contents

| 1. | Introduction | . 5 |
|----|---------------------------|-----|
| | Study Design | |
| 3. | Aims and Objectives | . 6 |
| 4. | Outcomes | . 6 |
| 5. | Population to be analyzed | . 6 |
| 6. | Analyses | . 6 |
| 7. | Missing data | . 6 |

Statistical Analysis Plan

**DORAGEN** 

1. Introduction

The aim of this project is to assess Doravirine concentrations in seminal plasma and

cervicovaginal fluid in HIV-1 infected male and female individuals receiving ART with

Doravirine plus TAF/FTC.

This statistical analysis plan (SAP) will give more detailed descriptions of the endpoints in the

study and the corresponding analyses.

2. Study Design

Study subjects will be selected from the routine control visits in the outpatient clinic of the HIV

and STD Unit at the Bellvitge University Hospital. Asymptomatic, HIV-1 infected individuals and

be on stable ART continuously or ≥3 consecutive months and Plasma HIV-1 RNA at <40

copies/mL for at least 3 months will be recruited.

This is Pilot study, Open label, single arm, single center, prospective study. Study patients will

receive one tablet of Doravirine 100 mg administered in combination with FTC and TAF

(Descovy®)).

Clinic visits will be performed at 3 time points: baseline, week 4 and week 8, only in baseline

and w8 HIV-1 RNA viral load and Doravirine cervicovaginal fluid and seminal plasma

concentration will be assessed.

2.1 Sample Size.

Fifteen male and fifteen female individuals will be included in the study. This is a study

designed to obtain information about doravirine concentrations and HIV viral suppression in

seminal plasma and cervicovaginal fluid. The study design is similar to other studies evaluating

PK and PD of antiretroviral drugs in these compartments.

# 3. Aims and Objectives

This study will address these unknowns and provide additional evidence for the scientific rational for the use of Doravirine in treatment and prevention strategies.

#### 4. Outcomes

- Concentration of Doravirine in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals, respectively, 8 weeks after switching to Doravirine plus TAF/FTC.
- HIV-1 RNA in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals, respectively, 8 weeks after switching to Doravirine plus TAF/FTC.

#### 4.1 Safety outcomes

#### **Adverse events**

Adverse events are reported at each clinic visit.

#### Concomitant medications

Usage of medications during study period will be recorded.

# 5. Population to be analyzed

## Per Protocol (PP)

All randomised study subjects completing the whole study period (complete cases). For a specific analysis, study subjects with missing data on any of the variables in the model will be excluded from the analysis.

# 6. Analyses

All outcomes will be presented using descriptive statistics; normally distributed data by the mean and standard deviation (SD) and skewed distributions by the median and interquartile range (IQR). Binary and categorical variables will be presented using counts and percentages.

The primary analysis will determine the Doravirine concentration in cervicovaginal fluid and seminal plasma and blood plasma, and the HIV-1 viral load in cervicovaginal fluid and seminal plasma and blood plasma.

# 7. Missing data

Subjects with missing data will be excluded for the analysis.